CLINICAL TRIAL: NCT03954990
Title: Treatment of Bacterial Vaginosis Prior to Active Labor and Infectious Morbidity: A Randomized Controlled Trial
Brief Title: Treatment of Bacterial Vaginosis Prior to Active Labor and Infectious Morbidity
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of significance/futile study
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-0103
Record Dates: First submitted 2019-04-23; First posted 2019-05-17 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Bacterial Vaginoses
Keywords: Bacterial Vaginoses in pregnancy
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Metronidazole

STUDY DESIGN:
Intervention Model Description: Patient with bacterial vaginosis will be randomized to either treatment group to receive 2 g of metronidazole or control group to receive 2 g of placebo. Randomization to either control or treatment group will be done according to a randomization sequence that is computer generated and maintained by investigational drug pharmacy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients, providers, PI, investigators will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control Arm (Placebo Comparator): Placebo tablets oral, 4 tablets once.
  Interventions: Drug: Placebo Oral Tablet
- Treatment Arm (Active Comparator): Will receive 4 tablets (2g) of metronidazole oral once.
  Interventions: Drug: Metronidazole Oral

INTERVENTIONS:
Drug: Metronidazole Oral — 4 tablets (2 g of metronidazole)
  Other Names: Flagyl
  Arms: Treatment Arm
Drug: Placebo Oral Tablet — 4 tablets
  Arms: Control Arm

SUMMARY:
Bacterial vaginosis (BV) is the most common cause of vaginal discharge among repro-ductive aged women. It is been linked to adverse maternal and neonatal outcomes. Our objective is to evaluate if the use of a single dose of metronidazole in women with BV at time of delivery reduces infectious morbidities

DETAILED DESCRIPTION:
The investigators are proposing a double-blinded, placebo controlled, randomized trial of 525 pregnant women undergoing induction or admitted in early labor and who are diagnosed with bacterial vaginosis. On admission to labor and delivery, patient will be counseled about the study. Patients who agree to be enrolled, will sign informed consent. Following enrollment patients will be screened for Bacterial vaginosis by doing a speculum exam and testing for Amsel's criteria. BV +ve patients will be randomized to receive either metronidazole 2 grams PO once or identically appearing placebo. The PI, study coordinator, or a collaborator will be responsible for the informed consent.

This will be a double-blinded randomized clinical trial. Neither the patient nor provider will be aware of treatment assignment. As with any other in-stance in which antibiotics are administered, there is a chance of an allergic or other adverse reaction. The patient will receive standard inpatient monitoring during the labor course and in the postpartum period, and so any immediate adverse reaction would be promptly detected.

Patient will be assessed intrapartum for development of chorioamninoitis. Postpartum patient will be assessed for infective complications up to 4 weeks. Neonates will be assessed for morbidities by chart review for 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Women ≤50 years at the time of admission with the ability to give informed con-sent.
* Admission for induction of labor or early spontaneous labor with cervix ≤3 cm.
* Diagnosed with bacterial vaginosis at time of admission or in the week prior to admission if not treated
* Gestational age ≥ 34 weeks

Exclusion Criteria:

* Spontaneous rupture of membranes
* Plan for elective cesarean delivery
* Allergy or contraindications to metronidazole
* Receipt of metronidazole or clindamycin in the admission for delivery for other in-dications.
* Hemodialysis
* Severe liver dysfunction
* Diagnosis of chorioamnionitis at the time of admission

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2022-09-26 (Actual)

PRIMARY OUTCOMES:
Rate of Composite outcome of maternal infections | Labor to 4 weeks postpartum
  Including Chorioamnionitis, postpartum endometritis, wound infection, pelvic septic thrombosis, pelvic or abdominal abscess

SECONDARY OUTCOMES:
Rate of Chorioamnionitis | From beginning of labor process until time of delivery
  Presumptive or confirmed diagnosis
Rate of Postpartum Endometritis | From time of delivery to 4 weeks postpartum
  Postpartum intrauterine infection
Rate of Surgical Site Infection | 4 weeks postpartum
  Including superficial or deep incisional surgical site infection
Rate of Pelvic Septic Thrombosis | 4 weeks postpartum
  Infection and thrombosis of pelvic vessels
Rate of Pelvic abscess | 4 weeks postpartum
  Detection of pelvic abscess on imaging
Rate of Puerperal fever | From beginning of labor process until time of delivery
  Temperature of ≥ 100.4 F at least twice 30 minutes apart or once ≥ 101F
Rate of Maternal Death | During labor and up to 4 weeks postpartum
  Death of mother while pregnant or within 28 days of pregnancy termination from any cause related to pregnancy or its management.
Rate of additional postpartum procedures | 4 weeks postpartum
  Additional imaging and invasive procedures to diagnose or treat postpartum infections
Rate of Postpartum Antibiotics use | 4 weeks postpartum
  Number of patients requiring antibiotics secondary to postpartum infections
Rate of ER and unscheduled postpartum clinic visit | 4 weeks postpartum
  Number of unscheduled clinic visits and ER visits secondary to infections.
Number of days of hospital stay postpartum | 4 weeks postpartum
  Number of days patients admitted to the hospital secondary to infections postpartum
Rate of Adverse events | 4 weeks postpartum
  Allergic reactions (anaphylaxis, angioedema, skin rashes including Stevens Johnson and Toxic Epidermal necrolysis), Gastrointestinal symptoms (nausea, vomiting, diarrhea, constipation, ileus, etc)
Rate of Confirmed neonatal sepsis | 7 days of delivery
  Findings indicating positive cultures of blood, cerebrospinal fluid or urine obtained by catheterization or suprapubic aspiration, or cardiovascular collapse, or an unequivocal X-ray confirming infection in a clinically septic neonate.
Rate of Suspected neonatal sepsis | 7 days of delivery
  Presence of clinical signs/symptoms (hypothermia, fever, irritability, poor feeding, hypotonia, etc) causing the clinician to perform a sepsis work-up (blood, urine and/or cerebrospinal fluid, or chest X-ray), excludes routine work-up solely for positive maternal Group B Streptococcus (GBS) status.
Rate of Neonatal morbidities | 90 days after delivery
  Including Respiratory Distress syndrome(RDS), Necrotizing enterocolitis(NEC), Intraventricular hemorrhage (IVH), Bronchopulmonary Dysplasia (BPD)

CONTACTS AND LOCATIONS:
Overall Officials: Sangeeta Jain, MD, Principal Investigator — University of Texas medical branch, Galveston
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States